## **COVER PAGE**

## **Inform Consent**

The Effect of Ophiocephalus striatus Extract on IGF-1 and IL-6

Levels in Elderly Patients with Sarcopenia

**Trial Registration Number:** NCT05869383

**Date of document:** 15 March 2023

| INFORMED CONSENT FORM IN RESEARCH | | |
|---|---|---|
| Researcher | dr. Nur Riviari, SpPD, K-Ger | |
| Information | dr. Nur Riviari, SpPD, K-Ger | |
| provider | | |
| Information | | Date |
| Type of | Content of Information | Mark |
| information Research title | The Effect of Ophiocephalus striatus Extract on IGF-1 and IL-6 Levels in Elderly Patients with Sarcopenia | |
| Research objectives | To determine the effect of Ophiocephalus striatus on IGF-1 and IL-6 levels in elderly patients with sarcopenia. | |
| Research methodology | Research Focus: This research is a clinical trial of a drug. Several aspects to be observed in this research include nutritional status measured through IGF-1 and IL-6 levels. Research Procedure: The research will be conducted at the Geriatrics and Internal Medicine Clinic, RSUP Dr. Mohammad Hoesin, Palembang. Interviews, physical examinations, and blood tests will be | |
| | conducted before and after the administration of the tested supplement to collect the required data. The physician will explain the background, purpose, and procedures of this clinical trial and inquire about the willingness to participate. If willing, participants will undergo subject selection involving | |
| | interviews, physical examinations, and laboratory tests (which may also refer to medical records). If the tests do not reveal significant liver and/or kidney function disorders, participants will be asked to consent to participate in this clinical trial. They will be given the tested supplement to consume for 2 weeks. After 2 weeks, participants will be re-interviewed, and blood samples will be taken again. | |

| Research risks | Participants may experience mild discomfort or pain during blood collection, occasionally accompanied by slight bruising, which will fade within a few days. Rarely, allergic reactions may occur. | |
|---|---|---|
| Research<br>benefits | By participating in this research, participants contribute valuable scientific information about the effects of Ophiocephalus striatus (snakehead fish) extract, particularly whether it can improve sarcopenia conditions in the elderly. | |
| Alternative procedures | There are no alternative procedures. | |
| Confidentiality of data | All information obtained during this research, including personal and research data, will be kept confidential. The participant's name or any documents identifying them as part of the research will not be disclosed without their consent. | |
| Compensation in case of side effects | Any significant incidents, such as hospitalization or death, must be reported to the researcher via phone. Participants experiencing complaints can contact the researcher 24/7 by phone. Participants reporting side effects will be asked to come for further anamnesis, physical examination, and laboratory tests as indicated. | |
| Researcher's Name and Address Number of | Dr. Nur Riviati, SpPD, K-Ger<br>Jl. DR. Hakim No. 1120, Sei Pangeran, Ilir<br>Timur I, Palembang | |
| subjects Potential hazards | Allergic reactions to Ophiocephalus striatus extract | |
| Cost incurred | In case of significant side effects | |
| Incentives for participants | Light refreshments | |
| I hereby state that I have explained the above matters truthfully and provided an opportunity for questions and/or discussions. | | Researcher's signature |
| I hereby state that I above, which I hav and I understand it. | Participant's signature | |